CLINICAL TRIAL: NCT06298214
Title: Testing the Effectiveness of the Her Health Program to Add Healthcare Value in the Fourth Trimester
Acronym: Her Health
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth F Sutton, PhD (Other)
Collaborators: Donaghue Medical Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Elizabeth F Sutton, PhD, Director of Scientific Research, Woman's
Organization: Woman's (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RP-23-019
Record Dates: First submitted 2024-02-08; First posted 2024-03-07 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Postpartum; Pregnancy Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Subjects will see doctors as normal during first year postpartum with no assistance.
- Her Health Program (Experimental): Her Health is a patient navigation intervention delivered by community health workers across the first postpartum year. Her Health has two interspersed components: Navigation and Education. Her Health Navigation is delivered through weekly and monthly check-ins between participant and navigator. Her Health navigators will deliver historically informed and culturally competent education designed to promote self-efficacy and self-advocacy within the healthcare system.
  Interventions: Behavioral: Her Health Program

INTERVENTIONS:
Behavioral: Her Health Program — Addition of a community health worker navigator to assist subject in navigating their health in the first year postpartum.
  Arms: Her Health Program

SUMMARY:
The goal of this clinical trial is to learn if a program Woman's Hospital has made, called the Her Health Program, can help women be healthy and get healthcare in the first year after having a baby.

The main question[s] the study aims to answer are:

* Can the Her Health program increase access to healthcare in the first year postpartum?
* Can the Her Health program increase knowledge about healthcare and change feelings toward the healthcare system?

Participants will complete one research visit in which they will be enrolled and told which group they will be in- "Her Health Program" group or "Usual Care" group. If they are placed in the "Her Health Program" group, they will receive their usual care + the addition of an extra healthcare team member(called a community health navigator) to to work with patients and care team for a year postpartum.

Researchers will compare those who receive the Her Health Program and those who do not receive the program to see if the Her Health Program can help women get healthcare in the first year after having a baby.

ELIGIBILITY:
Inclusion Criteria:

* At least 16 years old at the time of consent.
* Gave birth within 7 days before randomization
* Medicaid enrolled
* Address of residence within a disadvantaged area (ADI>5).
* Clearly understands the study procedures and visit schedule, alternative treatments, and risks involved with the study, and voluntarily agrees to participate by giving verbal and written informed consent

Exclusion Criteria:

* Use of private health insurance exclusively
* Does not speak English.
* Plans to move out of state during the study time period
* Unwilling to provide permission to link study records, medical records, and Medicaid and Vital Records Database records.
* Unwilling to provide informed consent
* Unwilling to be randomized.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum visit attendance | 12 weeks postpartum
  Visit attended between 6-12 weeks of delivery (yes/no)

SECONDARY OUTCOMES:
Medical trust | 12 months postpartum
  Group-Based Medical Mistrust Scale; scores range from 12-60 with higher scores indicating more mistrust
Health literacy | 12 months postpartum
  Rapid Estimate of Adult Literacy in Medicine (REALM); scores 0-66; higher score indicates high literacy
Self-efficacy | 12 months postpartum
  PROMIS General Self-Efficacy; scores range 5-50; higher score indicates higher self-efficacy
Healthcare costs | 12 months postpartum
  total cost of healthcare from Medicaid Claims Database within the first 12 months after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Sutton, PhD, Principal Investigator — Woman's Hospital, Louisiana
Locations (1):
- Woman's Hospital, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/14/NCT06298214/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-06): https://cdn.clinicaltrials.gov/large-docs/14/NCT06298214/ICF_001.pdf